CLINICAL TRIAL: NCT02887599
Title: Assessment of the Cytotoxic Immune Status of Pancreatic Cancer Patients and the Severity of the Cancer Using Measurement of Natural Killer Cell Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2016-0015
Record Dates: First submitted 2016-08-22; First posted 2016-09-02 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Group (Other): Pancreatic cancer patients
  Interventions: Procedure: Blood collection
- Control Group (Other): Healthy people without evidence of malignancy
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — 1ml of blood specimen collection

SUMMARY:
Pancreatic cancer is the 5th leading cause of cancer death and the worst prognostic cancer in the world. This is due to high recurrent rate after surgical resection and poor response to chemotherapy and radiotherapy.

Recent studies revealed that peri-tumoral structure and patients' immune status including cytotoxic immunity played significant role in the bad behavior of pancreatic cancer. While past studies focused on oncogenes and tumor suppressor genes, recent studies focused on patients' own immunity. Patients' immunity modified by cancer cells is found to be correlated to cancer progression and metastasis.

Natural killer cells, playing an important role in cytotoxic immune system, are revealed to be decreased in patients with lung cancer, ovarian cancer, prostate cancer, colorectal cancer, and breast cancer. And in melanoma mouse model, when NK cell was suppressed, cancer progression and metastasis were accelerated.

This study sought to find the correlation of patients' cytotoxic immune status to cancer progression and status by measurement of NK cell activity in pancreatic cancer patients. This would be basic support to construct a prognostic model of pancreatic cancer for early metastasis and post operational recurrence.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 and under 85
* Control group : incidental found benign pancreatic cyst, non-neoplastic gall bladder polyp (ex, cholesterol polyp), healthy people having no evidence of malignancy in check up within 1 year
* Patient group : histological diagnosed pancreatic cancer patients, clinically diagnosed pancreatic cancer patients by radiologic evaluation
* Agreed to enroll the study and signed informed consent

Exclusion Criteria:

* Patients with other malignancies within 5 years
* Patients treated with steroid due to any reason within 1 year
* Not signed informed consent

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Difference of the cytotoxic immune status | 24-hour after blood collection
  Difference of the cytotoxic immune status between patients group and control group by comparing quantitative measurements of NK cell activities by ELISA kit
Difference of the severity of the pancreatic cancer | 24-hour after blood collection
  Difference of the cytotoxic immune status according to the stage of the pancreatic cancer by comparing quantitative measurements of NK cell activities by ELISA kit

SECONDARY OUTCOMES:
Correlation of the cytotoxic immune status | 24-hour after blood collection
  Correlation of the cytotoxic immune status with tumor markers

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No